CLINICAL TRIAL: NCT01975493
Title: Neonatal and Paediatric Pharmacokinetics of Antimicrobials Study
Acronym: NAPPA
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: St George's, University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 13.0095; 2013-002366-40 (EudraCT Number); 13/LO/0907 (Other: Research Ethics Committee (REC))
Record Dates: First submitted 2013-09-23; First posted 2013-11-04 (Estimated); Last update posted 2018-03-21 (Actual); Status verified 2018-03

CONDITIONS: Paediatric Antimicrobial Pharmacokinetics
Keywords: Infectious Diseases; Paediatrics; Neonatology; Pharmacokinetics; Antimicrobials
MeSH Terms: conditions — Communicable Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Plasma samples and dried blood spots to be retained for retrospective analysis.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (6):
- Amoxicillin: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months) Children (2 - 11 years) Adolescents (12 - 16 years)
- Ampicillin: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months)
- Benzylpenicillin: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months) Children (2 - 11 years) Adolescents (12 - 16 years)
- Co-amoxiclav: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months) Children (2 - 11 years) Adolescents (12 - 16 years)
- Flucloxacillin: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months) Children (2 - 11 years) Adolescents (12 - 16 years)
- Piperacillin/tazobactam: Group subdivided into age categories:
  Preterm newborn infants Term newborn infants (0-27 days) Infants and toddlers (1 month to 23 months) Children (2 - 11 years) Adolescents (12 - 16 years)

SUMMARY:
The aim of NAPPA is to develop new models to improve our understanding of how children process ('metabolise') penicillins, to help us discover if we can improve the dosing regimens used for children in the future. The study population will involve children and neonates who need a penicillin antibiotic as part of their normal National Health Service (NHS) care, and who also need blood tests or intravenous access. Therefore the antibiotic study can be done without the need for any extra invasive procedures, and there will be no change to the medication therapy received by participants. In addition, NAPPA will evaluate whether it is feasible to measure antibiotic levels on a tiny drop of blood put onto absorbent paper ("dried blood spot"). This allows the sample to be stored and tested later on. NAPPA will compare the level of the antibiotic using this method with the level measured in the usual way, to show if this is a reliable method that could be used routinely in the future.

ELIGIBILITY:
Inclusion Criteria:

* Child aged under 16 years receiving one of the specified penicillins and with intravenous access or blood test(s) as part of their routine clinical care.
* Informed consent form signed by parent or legal guardian.

Exclusion Criteria:

* Any child or infant unlikely to survive 48 hours after recruitment.
* Patient known to be pregnant.
* Known allergy or hypersensitivity to beta-lactam antibiotics (including penicillins and cephalosporins) or beta-lactamase inhibitors.
* Patient receiving (or planned to receive) haemofiltration, haemodialysis, peritoneal dialysis, extracorporeal membrane oxygenation (ECMO) or cardiopulmonary bypass.

Ages: 1 Minute to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children (aged under 16 years) and infants (including both full-term and premature neonates), admitted to hospital and routinely prescribed one (or more) of the study penicillins according to local hospital policy.
Sampling Method: Non-Probability Sample
Enrollment: 428 (Actual)
Dates: Start 2013-11; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
The pharmacokinetic parameters of drug clearance and volume of distribution for each penicillin. | Participants will be followed for the duration of enrolment, an expected average of 7 days.

CONTACTS AND LOCATIONS:
Overall Officials: Mike Sharland, MD, Principal Investigator — St George's, University of London
Locations (9):
- United Kingdom (9):
  - Royal Cornwall Hospitals NHS Trust, Truro, Cornwall
  - Taunton and Somerset NHS Foundation Trust, Taunton, Somerset
  - University Hospitals Coventry and Warwickshire NHS Trust, Coventry
  - Alder Hey Children's Hospital, Liverpool
  - Liverpool Women's Hospital, Liverpool
  - St George's Hospital, London
  - Great Ormond Street Hospital, London
  - John Radcliffe Hospital, Oxford
  - Queen Alexandra Hospital, Portsmouth